CLINICAL TRIAL: NCT06106204
Title: A Parallel Cluster Randomized Trial of a Participatory Approach to Reduce Overuse of Antibiotics at Hospital Discharge: The ROAD Home Trial
Brief Title: Reducing Overuse of Antibiotics at Discharge Home
Acronym: ROAD Home
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Valerie Vaughn, Assistant Professor; Director of Hospital Medicine Research, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HS029482 (AHRQ)
Record Dates: First submitted 2023-10-07; First posted 2023-10-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia; Urinary Tract Infection; Antibiotic Stewardship; Care Transition
Keywords: Antibiotic Stewardship; Hospital Discharge; Urinary Tract Infection; Pneumonia; Facilitation; Adaptation; i-PARIHS Framework; Implementation Research Logic Model
MeSH Terms: conditions — Pneumonia; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel, cluster-randomized trial of 40 hospitals randomized to an implementation intervention designed to support antibiotic stewardship interventions vs. usual care control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROAD Home Intervention (Experimental): Hospitals randomized to receive the ROAD Home Intervention will receive an implementation intervention that includes external facilitation to support them in selecting and implementing evidence-based antibiotic stewardship strategies based on local context and the ROAD Home framework (https://academic.oup.com/cid/article/74/9/1696/6374407).
  Interventions: Other: ROAD Home Intervention
- Stewardship as Usual (No Intervention): Hospitals randomized to the control group will continue usual antibiotic stewardship activities. Although control hospitals are part of the HMS collaborative, during the intervention period they will not receive any of the ROAD Home Intervention components including analysis of their baseline data or needs assessment, customized suite of stewardship strategies, supported decision-making in selecting ROAD Home strategies to implement, an implementation blueprint, adaptable stewardship tools, or external facilitation from study investigators.

INTERVENTIONS:
Other: ROAD Home Intervention — Hospitals randomized to receive the ROAD Home Intervention will undergo (1) a baseline needs assessment to create a customized suite of stewardship strategies, (2) supported decision-making in selecting ROAD Home strategies to implement, and (3) external facilitation following an implementation blueprint.
  Arms: ROAD Home Intervention

SUMMARY:
The goal of this two-arm parallel cluster-randomized trial of 40 hospitals is to test the effectiveness of the ROAD Home Intervention on days of antibiotic overuse at discharge in patients hospitalized with community-acquired pneumonia (CAP) or urinary tract infection (UTI). The main question it aims to answer is: Does an antibiotic stewardship approach that is customized to the needs, goals, and resources of a hospital (i.e., the ROAD Home Intervention) compared to standard stewardship approaches reduce antibiotic overuse at discharge in hospitalized patients with CAP and UTI? The investigators will randomize 20 hospitals in the Michigan Hospital Medicine Safety Consortium (HMS) to the intervention group and 20 HMS hospitals to the "usual care" control group. During the study the investigators will: (a) assess baseline performance, existing stewardship strategies, hospital priorities, and resources; (b) develop a customized discharge stewardship "suite" for each intervention hospital based on the findings of the baseline assessment and informed by the ROAD Home Framework; and (c) support hospitals in selecting strategies and creating an implementation blueprint to be implemented over 12 to 15 months. After the intervention period, the investigators will compare days of antibiotic overuse at discharge and patient outcomes between intervention and "usual care" hospitals. It is hypothesized that hospitals randomized to the ROAD Home Intervention will have fewer days of antibiotic overuse at discharge compared to "stewardship as usual" control hospitals.

DETAILED DESCRIPTION:
The Reducing Overuse of Antibiotics at Discharge (ROAD) Home study is designed to test the hypothesis that hospitals randomized to an implementation intervention that includes external facilitation to support participants while allowing for free choice in selecting and implementing evidence-based antibiotic stewardship strategies based on local context will have fewer days of antibiotic overuse at discharge than "stewardship as usual" control hospitals. The first aim of this study is to evaluate the effectiveness of the ROAD Home Intervention on days of antibiotic overuse at discharge for hospitalized patients treated for CAP and UTI. The second aim of this study is to identify contextual factors influencing the implementation of the ROAD Home Intervention and to assess implementation outcomes (acceptability, feasibility, fidelity, and sustainment) to inform future broad dissemination.

A two-arm, parallel, cluster-randomized trial will assess the effect of the ROAD Home Intervention on days of antibiotic overuse at discharge. Forty hospitals will be recruited from the Michigan Hospital Medicine Safety Consortium (HMS; https://mi-hms.org/), a statewide 69-hospital collaborative consisting of diverse hospitals and focused on improving the care of hospitalized patients. HMS hospitals that agree to participate will undergo covariate-constrained randomization to improve balancing of critical hospital characteristics between groups with 1:1 allocation to the ROAD Home intervention vs. a "stewardship as usual" control. In the 12- to 15-month intervention period, hospitals will implement the intervention while investigators assess days of antibiotic overuse at discharge and patient outcomes. During the intervention period and in the 9-month post-intervention period, investigators will conduct a theory-informed mixed-methods process evaluation to evaluate barriers, facilitators, and implementation outcomes across hospitals.

ELIGIBILITY:
Inclusion Criteria:

All Patients:

* Adult patient admitted and discharged from the participating hospital and included in HMS registry
* Admitted to a general care medicine service
* Received any eligible antibiotic during the symptom collection window (-1 to +2 days for UTI; day 1 or 2 for pneumonia)
* Immunocompetent (allowing for mild immune suppression)
* Do not have a concomitant infection (e.g., antibiotic treatment for unrelated infection or prophylaxis)

Specific inclusion criteria for patients with UTI:

* Positive urine culture
* Have normal urinary anatomy

Specific inclusion criteria for patients with pneumonia:

- Discharge diagnosis of pneumonia

Exclusion Criteria:

All Patients:

* Left against medical advice or refused medical care
* Admitted on hospice
* Pregnant
* Unable to determine actual or expected antibiotic duration

Specific exclusions for patients with UTI:

- spinal cord injury

Specific exclusions for patients with pneumonia:

* Cystic fibrosis
* Pneumonia-related complication (e.g., empyema)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Days of antibiotic overuse at hospital discharge | 12 months; from discharge prescription
  Antibiotic overuse at discharge is a composite score of unnecessary antibiotic use, excessive antibiotic duration, and avoidable fluoroquinolones. The score is number of days of antibiotic overuse at hospital discharge.

SECONDARY OUTCOMES:
Number of cases with antibiotic-associated adverse events | 12 months; 30-days post hospital discharge
  This is a composite metric that includes patient-reported and physician-reported adverse events that are abstracted through chart review (routinely performed as part of being part of the HMS collaborative) as well as Clostridioides difficile laboratory events. The score is the number of cases who had antibiotic-associated adverse-events.

OTHER OUTCOMES:
Number of cases with composite 30-day outcome event | 12 months; 30-days post hospital discharge
  Composite 30-day outcome of mortality, readmission, and need for additional care (i.e., urgent/emergent visit) collected via patient phone call and chart review 30-days after hospital discharge. The score is the number of cases with a composite 30-day outcome event.
Number of cases with 30-day mortality | 12 months; 30-days post hospital discharge
  The score is the number of cases with 30-day outcome mortality.
Number of cases with 30-day readmission | 12 months; 30-days post hospital discharge
  The score is the number of cases with 30-day readmission.
Number of cases with 30-day C Difficile infection | 12 months; 30-days post hospital discharge
  The score is the number of cases with 30-day C Difficile infection.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie M Vaughn, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Hospitals enrolled in the study will report aggregate patient data. No IPD will be shared.

REFERENCES:
- [Background] Vaughn VM, Ratz D, Greene MT, Flanders SA, Gandhi TN, Petty LA, Huls S, Feng X, White AT, Hersh AL. Antibiotic Stewardship Strategies and Their Association With Antibiotic Overuse After Hospital Discharge: An Analysis of the Reducing Overuse of Antibiotics at Discharge (Road) Home Framework. Clin Infect Dis. 2022 Sep 29;75(6):1063-1072. doi: 10.1093/cid/ciac104. PMID 35143638
- [Background] Vaughn VM, Gandhi TN, Chopra V, Petty LA, Giesler DL, Malani AN, Bernstein SJ, Hsaiky LM, Pogue JM, Dumkow L, Ratz D, McLaughlin ES, Flanders SA. Antibiotic Overuse After Hospital Discharge: A Multi-hospital Cohort Study. Clin Infect Dis. 2021 Dec 6;73(11):e4499-e4506. doi: 10.1093/cid/ciaa1372. PMID 32918077
- [Background] Vaughn VM, Hersh AL, Spivak ES. Antibiotic Overuse and Stewardship at Hospital Discharge: The Reducing Overuse of Antibiotics at Discharge Home Framework. Clin Infect Dis. 2022 May 3;74(9):1696-1702. doi: 10.1093/cid/ciab842. PMID 34554249
- [Derived] Vaughn VM, Horowitz J, Gandhi T, Neetz RA, Petty L, Hersh A, Lindenauer P, Bernstein SJ, Flanders SA, Harrison JD, Smith JD, White AT, Szymczak JE. Developing an approach to enhance recruitment for a cluster-randomised implementation trial: leveraging deliberative participation and credible messengers. BMJ Open. 2025 Sep 16;15(9):e094925. doi: 10.1136/bmjopen-2024-094925. PMID 40962335
- [Derived] Szymczak JE, Petty LA, Gandhi TN, Neetz RA, Hersh A, Presson AP, Lindenauer PK, Bernstein SJ, Muller BM, White AT, Horowitz JK, Flanders SA, Smith JD, Vaughn VM. Protocol for a parallel cluster randomized trial of a participatory tailored approach to reduce overuse of antibiotics at hospital discharge: the ROAD home trial. Implement Sci. 2024 Mar 4;19(1):23. doi: 10.1186/s13012-024-01348-w. PMID 38439076
- See also: Michigan Hospital Medicine Safety Consortium Website — https://mi-hms.org/

DOCUMENTS (1):
  • Informed Consent Form (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT06106204/ICF_000.pdf